CLINICAL TRIAL: NCT01518413
Title: Phase 1 Dose Escalation Study of Sorafenib and Irinotecan Combination Therapy in Pediatric Patients With Relapsed or Refractory Solid Tumors
Brief Title: Dose Escalation Study of Sorafenib and Irinotecan Combination Therapy in Pediatric Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HMeany (Other)
Responsible Party: Sponsor-Investigator, HMeany, Holly Meany, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SorIrin1576
Record Dates: First submitted 2012-01-04; First posted 2012-01-26 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Rhabdomyosarcoma and Other Soft Tissue Sarcomas; Ewing's Sarcoma Family of Tumors; Osteosarcoma; Neuroblastoma; Brain Tumors
Keywords: Sora./Irino. combination therapy
MeSH Terms: conditions — Rhabdomyosarcoma; Osteosarcoma; Neuroblastoma; Brain Neoplasms | interventions — Sorafenib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Therapy (Experimental): Three to 6 patient will be enrolled at each dose level and dose escalations will proceed in the absence of dose-limiting toxicity attributed to therapy, first with dose escalation of sorafenib and then, if tolerated, escalation of irinotecan.
  Interventions: Drug: sorafenib; Drug: irinotecan

INTERVENTIONS:
Drug: sorafenib — sorafenib (50 and 200 mg tablets) orally twice daily, on a continuous schedule at a starting dose of 150mg/m2/dose.
Drug: irinotecan — irinotecan (70 mg/m2/dose) orally, concurrently, once daily,starting at the beginning of the 21 day cycle,repeated every 21 days

SUMMARY:
The purpose of this study is to determine the safest and most effective oral dose combinations of sorafenib and irinotecan in pediatric patients with solid tumors, i.e. relapsed or refractory.

DETAILED DESCRIPTION:
Sorafenib, a multi-kinase inhibitor of several targets felt to be important in tumor growth and angiogenesis, has been well studied and shown promising clinical results in adult cancer patients and the Maximum Tolerated Dose or MTD has been determined in pediatric patients. Irinotecan is known to be effective and is widely used in pediatric malignancies. The combination of sorafenib with irinotecan is of interest as these agents have different mechanisms of action. In addition, the combination has been evaluated in adult patients and deemed tolerable without alterations in the pharmacokinetic (PK) profile at the MTD. The trial we are proposing also offers the advantage of being a completely oral regimen, adding convenience and cost effectiveness. Given these considerations, if the sorafenib/irinotecan combination proves tolerable in phase I studies and shows efficacy in phase II studies, it would be an attractive combination to incorporate into existing chemotherapy regimens for pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

* AGE: >=2 year and <22 years of age.

  * DIAGNOSIS: solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing's sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilms' tumor, hepatic tumors, germ cell tumors and brain tumors.
  * MEASURABLE/EVALUABLE DISEASE: Patients must have measurable or evaluable disease.
  * THERAPEUTIC OPTIONS:
* The patient's cancer must have relapsed after or failed to respond to frontline curative therapy and there must not be other potentially curative treatment options available. Curative therapy may include surgery, radiation therapy, chemotherapy, or any combination of these modalities.

  • PRIOR THERAPY:
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to enrolling on this study.
* No limitation on the number of prior chemotherapy regimens that the patient may have received prior to study enrollment.
* Myelosuppressive chemotherapy: The last dose of all myelosuppressive anticancer drugs must be at least 3 weeks prior to study entry.
* Immunotherapy: The last dose of immunotherapy (monoclonal antibody or vaccine) must be at least 4 weeks prior to study entry.
* Biologic (anti-cancer agent): The last dose of all biologic agents for the treatment of the patient's cancer (such as retinoids or tyrosine kinase inhibitors) must be at least 7 days prior to study entry. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Investigational anti-cancer agent: The last dose of all investigational agents must be at least 30 days prior to study entry.
* Radiation therapy: The last dose of radiation to more than 25% of marrow containing bones (pelvis, spine, skull) must be at least 4 weeks prior to study entry. The last dose of all other local palliative (limited port) radiation must be at least 2 weeks prior to study entry.
* Stem Cell Transplantation. At least 2 months post-autologous stem cell transplant or at least 3 months post-allogeneic transplant and recovered from toxicities without evidence of graft versus host disease.
* Prior camptothecins: Patients who previously received irinotecan as front line treatment or in an adjuvant setting are eligible if they did not experience severe toxicities (defined as grade 4 non-hematologic toxicity or failure to recover from any non-hematologic or hematologic toxicity within 6 weeks of receiving the drug) possibly, probably or definitely related to the agent, and they did not experience tumor progression during the time they received the agent. Patients who previously received topotecan are eligible.
* Growth Factors. The last dose of colony stimulating factors, such as filgrastim, sargramostim, and erythropoietin, must be at least 1 week prior to study entry, the last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be at least 2 weeks prior to study entry.

  • CONCURRENT THERAPIES:
* No other anti-cancer therapy (chemotherapy, biological therapy, radiation therapy) is permitted.

  • PERFORMANCE STATUS:
* Patients > 10 years old must have a Karnofsky performance level >= 50%, and children <= 10 years old must have a Lansky performance level >= 50%.
* Patients who are unable to walk because of paralysis or motor weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.

  • HEMATOLOGIC FUNCTION:
* Peripheral absolute neutrophil count (ANC) of >=750/mcL
* Platelet count >=75,000/mcL without administration of platelets

  • HEPATIC FUNCTION:
* Total bilirubin must be gender
* SGPT (ALT) must be - Serum albumin >/= 2 g/dL

  * RENAL FUNCTION: Age-adjusted normal serum creatinine (see table below) OR a creatinine clearance >=60 mL/min/1.73 m2. Age Maximum Serum Creatinine (Years) (mg/dl) Male Female 2 to less than 6 years 0.8 0.8 6 to less than 10 years 1 1 10 to less than 13 years 1.2 1.2 13 years to less than 16 years 1.5 1.4 Greater than or equal to 16 years 1.7 1.4 The threshold creatinine values in this table were derived from the Schwartz formula for estimating GFR (Schwartz et.al. J Peds 106:522, 1985) utilizing child length and stature data published by the CDC.
  * ADEQUATE PULMONARY FUNCTION: Defined as no dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air if there is clinical indication for determination (cough, etc).
  * Normal serum amylase and lipase
  * PT and PTT <= 1.5 times the upper limit of normal for age (including patients on prophylactic anticoagulation). Prophylactic anticoagulation as described below is permitted:
  * Low dose warfarin with PT-INR <= 1.5 x ULN. For subjects receiving warfarin, the PT-INR should be measured prior to initiation of trial drugs and should be monitored at least weekly, or as defined by the local standard of care, until it is stable.
  * Low-dose aspirin (<= 100 mg daily).
  * Prophylactic doses of heparin.
  * Blood pressure (BP) <= the 95th percentile for age, height and gender and not receiving anti-hypertensive medications or well controlled on antihypertensive medications for one week. Blood pressure will be recorded as the average of 2 measurements separated by at least 2 minutes. If the second value is more than 5 mmHg different from the first, continued measurements should be made every 2 minutes until a stable value is attained. The recorded value should be the average of the last two measurements obtained. Blood pressure is to be measured preferably in the right arm with an appropriate sized cuff, taken in a seated position after 3 minutes of rest. Oscillometric blood pressure measurements that exceed the 95th percentile should be confirmed by auscultation.
  * BIRTH CONTROL: Patients of childbearing or child-fathering potential will be required and must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

Exclusion Criteria:

* Clinically significant unrelated systemic illness, such as serious infections, hepatic,renal or other organ dysfunction, which in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate the agents used in this trial or are likely to interfere with the study procedures or results.

  * Patients with known intra-axial metastatic central nervous system lesions.
  * Pregnant or breast-feeding females are excluded because of the potential harmful effects of sorafenib and irinotecan on a developing fetus or nursing child.
  * Patients currently receiving other anticancer agents or radiation therapy.
  * Patients currently receiving other investigational agents.
  * Prior treatment with a sorafenib containing regimen.
  * Inability to swallow pills.
  * Evidence of bleeding diathesis and/or on therapeutic anti-coagulation medications.
  * Patients with known Gilbert syndrome.
  * Patients who take cytochrome P450 enzyme-inducing antiepileptic agents (phenytoin, carbamazepine, phenobarbitol), rifampin, erythromycin, azithromycin, azole antifungals, grape fruit juice or St. Johns Wort. Patients must have discontinued these medications at least 7 days prior to enrollment of trial.
  * Patients with baseline hypertension (>=95th BP percentile for age, height and gender) and not controlled on anti-hypertensive medications.
  * Patients with a malabsorption syndrome.
  * Patients with known human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection.
  * Patients with serious non-healing wound, ulcer, or bone fracture.
  * Patients with thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
  * Patients with cardiac ventricular arrhythmias requiring anti-arrhythmic therapy,unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
  * Patients who have undergone major surgery, open biopsy or significant traumatic injury within 4 weeks of study enrollment.
  * Patients with known or suspected allergy to any agent given in the course of this trial.

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2011-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Toxicity Profile | 24 months
  Determine the toxicity profile, dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of sorafenib, when administered in combination with oral irinotecan in children with relapsed or refractory solid tumors.
Patient Related Outcomes | 24 months
  Demonstrate the feasibility of incorporating measurement of patient-related outcome into a four site phase 1 trial of sorafenib and irinotecan for children and adolescents.
  Demonstrate feasibility: defined as 70% of participants will complete the 5 patient-reported outcomes (PROs) (pain, fatigue, worry, sadness and physical functioning) at both baseline (pre-treatment) and at the end of the first course and missing data will not be greater than 15% across the 5 PROs at either data point.

SECONDARY OUTCOMES:
Pharmacokinetic Profile | 24 months
  Describe the plasma pharmacokinetic profile of sorafenib and irinotecan when administered as combination therapy in children and adolescents.
Disease Evaluation | 24 months
  Evaluate disease response, based on criteria for measurable lesions (RECIST) and evaluable lesions, to guide further development in phase 2 studies.
Integration of Patient Related Outcomes with other outcome measures | 24 months
  Correlate and integrate the PRO scores with traditional endpoints of toxicity, pharmacokinetic profile, and tumor response associated with the sorafenib and irinotecan combination.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Meany, MD, Principal Investigator — Children's National Research Institute
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - National Cancer Institute, Bethesda, Maryland
  - Children's Hospital Boston/Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Meany HJ, Widemann BC, Hinds PS, Bagatell R, Shusterman S, Stern E, Jayaprakash N, Peer CJ, Figg WD, Hall OM, Sissung TM, Kim A, Fox E, London WB, Rodriguez-Galindo C, Minturn JE, Dome JS. Phase 1 study of sorafenib and irinotecan in pediatric patients with relapsed or refractory solid tumors. Pediatr Blood Cancer. 2021 Nov;68(11):e29282. doi: 10.1002/pbc.29282. Epub 2021 Aug 12. PMID 34383370